CLINICAL TRIAL: NCT05242510
Title: Divergence Excess/Simulated Divergence Excess Exotropia (DESDEE)
Brief Title: Evaluation of Exotropia After Patching the Eye or After Prism Adaptation
Acronym: DESDEE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of ability to enroll from other sites
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Matthew Gearinger, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006849
Record Dates: First submitted 2022-01-24; First posted 2022-02-16 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Exotropia
MeSH Terms: conditions — Exotropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patching (Experimental)
  Interventions: Procedure: Patching
- Prism Adaptation (Experimental)
  Interventions: Procedure: Prism Adaptation

INTERVENTIONS:
Procedure: Patching — The subject will occlude the non-dominant eye for 24 hours.
  Arms: Patching
Procedure: Prism Adaptation — The subject will undergo prism adaptation targeting the pre-occlusion distance angle for 1-2 weeks. • Fresnel prism(s) will be applied to the patient's spectacles equaling the distance angle between the two eyes. At the examiner's discretion depending on the size of the deviation, the prism(s) can be placed solely over the non-dominant eye, or split between the 2 eyes in some combination which results in equalization of the distance exotropia. If the distance angle calls for an amount of prism that cannot be exactly replicated with Fresnel prisms (e.g., 32 PD), the amount of prism used will be determined by rounding down to the nearest practical amount at examiner discretion.
  Arms: Prism Adaptation

SUMMARY:
This study intends to determine the number and percent of subjects initially diagnosed with divergence excess exotropia which would be reclassified as simulated divergence excess exotropia if tested after 24 hours of monocular occlusion (patching) or after prism adaptation for the distance angle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with divergence excess exotropia according to standard criteria (see Study Procedures for specifics)
* No prior strabismus surgery
* Able to cooperate with testing (by examiner determination)
* Neurologically normal except for strabismus (ADHD and autism spectrum are not exclusion criteria as long as the subject can cooperate for necessary testing)
* Not amblyopic at the time of enrollment (best-corrected visual acuity in both eyes of 20/40 or better)
* Under 18 years of age. There is no lower age limit as long as the subject can cooperate for the required testing.
* No diagnosis of dissociated vertical deviation

Exclusion Criteria:

* No diagnosis of divergence excess exotropia according to standard criteria (see Study Procedures for specifics)
* Prior strabismus surgery
* Unable to cooperate with testing (by examiner determination)
* Diagnosed with a neurological disorder (ADHD and autism spectrum are not exclusion criteria as long as the subject can cooperate for necessary testing)
* Best-corrected visual acuity in either eye worse than 20/40
* 18 years of age or older
* Diagnosed with dissociated vertical deviation

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Percent of participants reclassified as divergence excess exotropia | 2 weeks
  Percentage of patients with distance and near exotropia measurements within 2.5 prism diopters on alternate prism and cover testing after 24 hours of patching or 7-14 days of fresnel prism use.
Percent of participants reclassified as simulated divergence excess exotropia | 2 weeks
  Percentage of patients with distance and near exotropia measurements differing by more than 2.5 prism diopters on alternate prism and cover testing after 24 hours of patching or 7-14 days of fresnel prism use.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - University of California Los Angeles, Los Angeles, California
  - Harvard University, Boston, Massachusetts
  - Ross Eye Institute, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Queen's University, Kingston, Ontario, Canada
- LV Prasad Eye Institute, Hyderabad, India
- Shamir Medical Center, Rishon LeZiyyon, Central District, Israel
- University of Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No